CLINICAL TRIAL: NCT02765594
Title: Hydroxychloroquine Sulfate Alleviates Persistent Proteinuria in IgA Nephropathy:a Single Center Prospective Randomized Controlled Study
Brief Title: Hydroxychloroquine Sulfate Alleviates Persistent Proteinuria in IgA Nephropathy
Acronym: HCQIgAN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCHHCQIgAN01
Record Dates: First submitted 2016-04-30; First posted 2016-05-06 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Primary IgA Nephropathy
Keywords: Glomerulonephritis, IGA; Kidney Diseases; Autoimmune Diseases; Glomerulonephritis; Nephritis; Immune System Diseases; Urologic Diseases; Hydroxychloroquine; Anti-Infective Agents; Antimalarials; Antiparasitic Agents; Antiprotozoal Agents; Antirheumatic Agents; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action; Pharmacologic Actions; Therapeutic Uses; interleukin-6; interferon-alpha; tumor necrosis factor-alpha
MeSH Terms: conditions — Glomerulonephritis, IGA; Kidney Diseases; Autoimmune Diseases; Glomerulonephritis; Nephritis; Immune System Diseases; Urologic Diseases | interventions — Hydroxychloroquine; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- valsartan only:control group (Experimental): valsartan (160mg/d)
  Interventions: Drug: Valsartan
- hydroxychloroquine with valsartan:study group (Experimental): valsartan (160mg/d) and Hydroxychloroquine Sulfate ( 400mg/d, twice daily)
  Interventions: Drug: Hydroxychloroquine Sulfate; Drug: Valsartan

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate — 200mg bid
  Other Names: Fenle
  Arms: hydroxychloroquine with valsartan:study group
Drug: Valsartan — 160mg qd
  Other Names: Diovan

SUMMARY:
Immunoglobulin A nephropathy (IgAN) is the most common primary glomerulonephritis in the world.There is to date no curative therapy for patients with IgAN.It is considered that dendritic cells, Toll-like receptor (TLR) 9 and cytokines interleukin-6 (IL-6), and interferon-alpha (IFN-a) and tumor necrosis factor-alpha (TNF-α), play an important role in the aberrant mucosal response. Hydroxychloroquine is an antimalarial agent and had a notable impact on immune activation by the reduction of circulating activated immune cells that including decreased TLR-expressing cells, reduced IFN-secreting plasmacytoid dendritic cells, reduced production of inflammatory cytokines including interferon alpha, IL-6 and TNF alpha. Recent studies showed hydroxychloroquine had a benefit for renal remission and could retard the onset of renal damage in patients with lupus nephritis. hydroxychloroquine may have the potential effect in IgA nephropathy, alleviated the proteinuria and had the renal protect effect. This will be a single center, prospective, randomized, controlled study to assess the utility of hydroxychloroquine in IgAN patients.

DETAILED DESCRIPTION:
Immunoglobulin A nephropathy (IgAN) is the most common primary glomerulonephritis in the world. Its estimated frequency is at least 2.5 cases per year per 100,000 adults. The glomerulopathy usually progressed slowly leading to end stage renal disease (ESRD). ESRD developed in 20%-40% of patients after 20 years. Given its complex and as yet incompletely understood pathogenetic mechanisms, there is to date no curative therapy for patients with IgAN.

Although pathogenesis of IgAN is still obscure, underglycosylated IgA-containing immune-complex including IgG or IgA antibodies against the hinge region of IgA1 are key factors for IgA nephropathy. Aberrant mucosal immune response might lead to increased production of underglycosylated IgA1. It is considered that dendritic cells, Toll-like receptor (TLR)9, and cytokines interleukin-6 (IL-6), , interferon-alpha (IFN-a) and tumor necrosis factor-alpha (TNF-α), play an important role in the aberrant mucosal response.

Hydroxychloroquine is an antimalarial agent and had a notable impact on immune activation by the reduction of circulating activated immune cells that including decreased TLR-expressing cells, reduced IFN-secreting plasmacytoid dendritic cells, reduced production of inflammatory cytokines including interferon alpha, IL-6 and TNF alpha. Recent studies showed hydroxychloroquine had a benefit for renal remission and could retard the onset of renal damage in patients with lupus nephritis.

Therefore, hydroxychloroquine, targeting dendritic cells, TLR, IL-6, IFN-α and TNF-α，may have the potential effect in IgA nephropathy, alleviated the proteinuria and had the renal protect effect. This will be a single center, prospective, randomized, controlled study to assess the utility of hydroxychloroquine added to valsartan in IgAN patients.

ELIGIBILITY:
Inclusion Criteria:

1. biopsy proven primary IgA nephropathy
2. age 18-60 years
3. proteinuria range from 0.5 to 1.5g/d
4. serum creatinine ≤132.6μmol/L
5. normal blood pressure or blood pressure ≤130/80 mmHg in patients with hypertension

Exclusion Criteria:

1. Hypersensitivity to chloroquine or to hydroxychloroquine
2. blood pressure <90/60 mm Hg
3. pregnancy and breastfeeding women
4. renal artery stenosis
5. Rapidly progressive renal insufficiency
6. systemic lupus erythematosus or other connective tissue diseases
7. Henoch- schoenlein purpura
8. other nephritis
9. diabetes mellitus
10. retinopathy
11. other contraindication of hydroxychloroquine
12. severe hepatic insufficiency
13. G6PD deficiency
14. psoriasis or porphyria
15. malignant hypertension
16. viral hepatitis or other infections
17. treatment with steroids or cytotoxic drugs during the previous three months
18. psychiatric disorder
19. not suitable for the study judged by investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Remission (Complete [CR] or Partial [PR]) at Week 24 | 24 weeks
  CR: proteinuria <0.3 g/24 hr with no worsening of renal function (<15% estimated glomerular filtration rate(eGFR) reduction from Baseline).PR: proteinuria <3.5g/24 hrs but ≥0.3g/24 hrs and a decrease of >50% from Baseline based on 24 hours pooled urine, with no worsening of renal function(<15% eGFR reduction from Baseline). eGFR at Baseline will be defined as the Day 0 values.

SECONDARY OUTCOMES:
Change from Baseline in Proteinuria Levels at the Indicated Time Points | Baseline and Weeks 4, 12, 24
  Proteinuria is being assessed at Weeks 0, 4, 12, 24 follow-up visits. Proteinuria is based on 24 hours pooled urine. Baseline is defined as the Day 0 values. The ratio is defined as the post-Baseline value divided by the Baseline value.
Change from Baseline in Serum Creatinine Levels at the Indicated Time Points | Baseline and Weeks 4, 12, 24
  Serum creatinine is being assessed at Weeks 0, 4, 12, 24 follow-up visits. Baseline is defined as the Day 0 values. The ratio is defined as the post-Baseline value divided by the Baseline value.
Change from Baseline in eGFR at the Indicated Time Points | Baseline and Weeks 4, 12, 24
  eGFR is being assessed from levels of creatinine using the 4 variable version of the modification of diet in renal disease (MDRD) equation as recommended by national kidney foundation-chronic kidney disease (NKF-CKD) guidelines. eGFR is calculated at Weeks 0, 4, 12, 24 follow-up visits. Baseline is defined as the Day 0 values. The ratio is defined as the post-Baseline value divided by the Baseline value.
Change from Baseline in Serum IgA Levels at the Indicated Time Points | Baseline and Weeks 4, 12, 24
  IgA levels in serum are being analyzed at Weeks 0, 4, 12, 24 follow-up visits. Baseline is defined as the Day 0 value. The ratio is defined as the post-Baseline value divided by the Baseline value.
Change from Baseline in Serum Interleukin-6 Levels at the Indicated Time Points | Baseline and Weeks 4, 12, 24
  Interleukin-6 levels in serum are being analyzed at Weeks 0, 4, 12, 24 follow-up visits by means of enzyme linked immunosorbent assay (ELISA). Baseline is defined as the Day 0 value. The ratio is defined as the post-Baseline value divided by the Baseline value.
Change from Baseline in Serum Interferon alfa Levels at the Indicated Time Points | Baseline and Weeks 4, 12, 24
  Interferon alfa levels in serum are being analyzed at Weeks 0, 4, 12, 24 follow-up visits by means of enzyme linked immunosorbent assay (ELISA). Baseline is defined as the Day 0 value. The ratio is defined as the post-Baseline value divided by the Baseline value.
Change from Baseline in Serum Tumor Necrosis Factor alpha Levels at the Indicated Time Points | Baseline and Weeks 4, 12, 24
  Tumor necrosis factor alpha levels in serum are being analyzed at Weeks 0, 4, 12, 24 follow-up visits by means of enzyme linked immunosorbent assay (ELISA). Baseline is defined as the Day 0 value. The ratio is defined as the post-Baseline value divided by the Baseline value.
Adverse Effects at the Indicated Time Points | Weeks 4, 12, 24

CONTACTS AND LOCATIONS:
Overall Officials: RUITONG GAO, MD, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peing Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639